CLINICAL TRIAL: NCT02839369
Title: The Effect of Changing Walking Conditions on Walking Dynamic Characteristics Among Children Post a Severe Traumatic Brain Injury, Cerebral Palsy and Typically Developed (TD) Control.
Brief Title: Walking Dynamic Among Children With Brain Damge
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 158-08
Record Dates: First submitted 2010-02-28; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Traumatic Brain Injury; Cerebral Palsy
Keywords: walking performance; Cerebral Palsy, Typically Developed
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Palsy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children: post Traumatic Brain Injury With Cerebral Palsy Typically developed
  Interventions: Other: walking under varies conditions

INTERVENTIONS:
Other: walking under varies conditions — The children were asked to walk an electronic mat, three cycles for each one of the different trials as comfortable regular speed, walking as fast and as slow as possible, walking on straight line etc
Other: walking under varies conditions — walking on electronic walkway under different conditions

SUMMARY:
The goal of the present study was to look at the effect of changing walking parameters on the dynamic walking characteristics among children post severe traumatic brain injury, children with cerebral palsy and typically developed controls.

DETAILED DESCRIPTION:
leisure time physical activity by the Godin and Shephard (G&S) questionnaire. Balance tests - the Timed Up and Go test (TUG) and functional reach test (FRT). Maximal isometric strength was assessed by using a hand held dynamometer; walking dynamics were recorded by an electronic mat, and the 6 minute walk test, energy expenditure index (EEI) and perceived exertion by the OMNI scale.

ELIGIBILITY:
Inclusion Criteria:

Post Traumatic Brain Injury

* Post severe closed head injury (Glasgow Coma Scale (GCS) score at admission to emergency room of ≤8
* At least one year post trauma
* Ages 7 to 13 years
* Independent ambulation (foot orthoses permitted)

Children with Cerebral palsy

* GMFCS 1 or 2
* Ages 7 to 13 years
* Able to stand up from a chair independently and maintain standing for more than 5 seconds without falling, without obvious limitation in the passive range of motion of lower extremities.

Typically Developed age and sex controls exclusion criteria:

* Children who could not fulfill simple instructions

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children post Traumatic Brain Injury with Cerebral palsy Typically Developed
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
step characteristics | 30 minutes
  The Gaitrite system - step length and time variability (%).

SECONDARY OUTCOMES:
step time | part of the first assessment
  step time in sec
step length | part of the first assessment
  step length in cm
gait velocity | part of the first assessment
  walking velocity (cm/sec),

CONTACTS AND LOCATIONS:
Locations (1):
- Alyn Children's Rehabilitation Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No